CLINICAL TRIAL: NCT05418530
Title: Effect of Closed Tracheal Aspiration Associated With Expiratory Pause in Pediatrics: A Randomized, Crossover Clinical Study
Brief Title: Effect of Closed Tracheal Aspiration Associated With Expiratory Pause in Pediatrics Randomized, Crossover Clinical Study
Acronym: expirapause
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: expiratory pause_2022
Record Dates: First submitted 2022-03-03; First posted 2022-06-14 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-03

CONDITIONS: Respiratory Insufficiency in Children
Keywords: Respiratory Insufficiency, respiratory artificial
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: Patients who meet the inclusion criteria and after signing the informed consent by the guardian will be randomized to closed system aspiration with an expiratory pause and closed system aspiration without an expiratory pause. Randomization will be performed by blocks of sealed envelopes, allocating the patient to a first technique to be performed and, after 6 hours, to another technique. All patients will perform both forms of aspiration and will be aspirated 2 hours before the start of each technique to match the groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- with pause- without pause (Active Comparator): Start with an expiratory pause during aspiration and after 6hours the aspiration is performed without an expiratory pause
  Interventions: Other: with pause- without pause
- without pause - with pause (Active Comparator): Start without an expiratory pause during aspiration and after 6hours the aspiration is performed with an expiratory pause
  Interventions: Other: without pause-with pause

INTERVENTIONS:
Other: with pause- without pause — start with pause expiration
  Arms: with pause- without pause
Other: without pause-with pause — start without pause expiration
  Arms: without pause - with pause

SUMMARY:
Introduction: Patients on mechanical ventilation suffer alterations in the viscoelastic characteristics of the mucus due to changes in the humidity and temperature of the inhaled air and in the respiratory volumes and flows. The literature has pointed out the use of mechanical ventilators as a tool for mobilizing secretions and closed-system aspiration associated with expiratory pause has been shown to be effective in mobilizing secretions. Objectives: To assess whether there is a difference in the mass of aspirated secretion with the application of the expiratory pause during aspiration. Methods: A crossover, randomized study. Applied to children aged 0 to 5 years and 11 months who are intubated for 24 hours with orotracheal tubes or tracheostomy. There will be an exclusion of patients who present with undrained pneumothorax, cranial hypertension or any other clinical situation that has a clinical contraindication to aspiration and patients whose parents do not agree to participate in the study. The technique will be during aspiration in the tube with where to apply or not the expiratory pause on the mechanical ventilator. This secretion will be weighed so that there is fidelity in the results.

DETAILED DESCRIPTION:
A prospective, crossover, randomized clinical study will be carried out in the Pediatric ICU of Hospital Israelite Albert Einstein.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 0 to 5 years and 11 months who have been on invasive mechanical ventilation for more than 24 hours through an orotracheal cannula or tracheostomy will be included in the study.

Exclusion Criteria:

* Patients who present with undrained pneumothorax, cranial hypertension or any other clinical situation that has a clinical contraindication to aspiration and patients whose parents do not agree to participate in the study will be excluded from the study.

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2022-04-22 (Actual); Primary Completion 2022-04-22 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
secretion mass | 6 hours
  The secretion will be weighed on a scale graduated in milligrams.

SECONDARY OUTCOMES:
tidal volume | 6 hours
  tidal volume checked on the mechanical ventilator graduated in ml

CONTACTS AND LOCATIONS:
Locations (1):
- Albert Eisntein Hospital, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
the results of the study can be requested by the person responsible for the patient and these will be sent by emial